CLINICAL TRIAL: NCT03087474
Title: Treatment of Venous Thromboembolism in Real-Life Patients: A Nationwide, Population-Based Study
Brief Title: Treatment of Venous Thromboembolism in Real-Life Patients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-496
Record Dates: First submitted 2017-03-02; First posted 2017-03-22 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VKA patients: Vitamin K antagonist (VKA) patients
  Interventions: Other: Non-Interventional
- NOAC patients: nonvitamin K antagonist oral anticoagulants (NOAC) patients
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
In a population of patients with venous thromboembolism and treated with oral anticoagulants (OAC) in routine clinical practice in Denmark this study will describe patients treated with each OAC

ELIGIBILITY:
Inclusion Criteria:

1. All patients ≥ 18 years diagnosed with incident VTE at Danish public hospitals from 2006 through 2015
2. First-time (index) VTE will be defined as an in- or out-patient diagnosis of DVT or PE among patients redeeming a prescription for anticoagulant drugs within 30 days after index date

Exclusion Criteria:

1. In the analyses on type and duration of anticoagulant use, Patients with cancer will be excluded as they typically receive low molecular heparin directly from the hospital and their use of anticoagulants can therefore not be captured by redeemed prescriptions at pharmacies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Danish National Patient Registry (DNPR), covering all Danish hospitals, will be used to identify first-time and recurrent VTE cases diagnosed from 01-Jan-2006 through 31-Dec-2015.
Sampling Method: Non-Probability Sample
Enrollment: 89383 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate in VKA patients for VTE | Approximately 180 months
  Hospitalization rate for first-time Venous thromboembolism (VTE) in Vitamin K antagonist (VKA) patients
VTE hospitalization rate in VKA patients by sex | Approximately 180 months
VTE hospitalization rate in VKA patients by age | Approximately 180 months
Hospitalization rate in NOAC patients for VTE | Approximately 180 months
  Hospitalization rate for first-time venous thromboembolism in nonvitamin K antagonist oral anticoagulants (NOAC) patients
VTE hospitalization rate in NOAC patients by sex | Approximately 180 months
VTE hospitalization rate in NOAC patients by age | Approximately 180 months
Duration of Treatment in NOAC patients | Approximately 180 months
Duration of treatment in VKA patients | Approximately 180 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx